CLINICAL TRIAL: NCT05283642
Title: The Effects of D-chiro-inositol in Endometrial Thickness
Brief Title: D-chiro-inositol and Endometrial Thickness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lo.Li.Pharma s.r.l (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: DCI_GYN22
Record Dates: First submitted 2022-03-08; First posted 2022-03-17 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-03

CONDITIONS: Endometrial Diseases
MeSH Terms: conditions — Uterine Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DCI (Experimental): Oral supplementation with D-chiro-inositol once a day
  Interventions: Dietary Supplement: DCI

INTERVENTIONS:
Dietary Supplement: DCI — Oral supplementation with D-chiro-inositol once daily

SUMMARY:
Investigation of the effects of D-chiro-inositol supplementation in women with altered endometrial thickness.

ELIGIBILITY:
Inclusion Criteria:

- altered endometrial thickness

Exclusion Criteria:

* patients with cancer
* patients under hormonal treatments (progestogens and/or estrogens)
* patients supplemented with inositols

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2022-03-08 (Actual); Primary Completion 2022-10-29 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Change in endometrial thickness | Two time points: baseline and after three months
  Change in endometrial thickness by ultrasound measurement from baseline to three months

CONTACTS AND LOCATIONS:
Locations (1):
- ASL Umbria 2, Terni, Umbria, Italy